CLINICAL TRIAL: NCT04933188
Title: Early Detection of Myocardial Work Impairment in Patients With Overweight and Obesity (EARLY-MYO-OBESITY-II)
Brief Title: Early Detection of Myocardial Work Impairment in Obesity II(EARLY-MYO-OBESITY-II)
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Ningbo Hangzhou Bay Hospital (Unknown); Jiading Central Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: ACFO2020
Record Dates: First submitted 2021-03-30; First posted 2021-06-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: Lean health controls with a BMI<25kg/m2
  Interventions: Diagnostic Test: Myocardial work was estimated from left ventricular pressure-strain loop derived from speckle tracking echocardiography and non-invasive brachial artery cuff pressure
- overweight: patients with a BMI of 25-30kg/m2
  Interventions: Diagnostic Test: Myocardial work was estimated from left ventricular pressure-strain loop derived from speckle tracking echocardiography and non-invasive brachial artery cuff pressure
- obesity: patients with a BMI of over 30kg/m2
  Interventions: Diagnostic Test: Myocardial work was estimated from left ventricular pressure-strain loop derived from speckle tracking echocardiography and non-invasive brachial artery cuff pressure

INTERVENTIONS:
Diagnostic Test: Myocardial work was estimated from left ventricular pressure-strain loop derived from speckle tracking echocardiography and non-invasive brachial artery cuff pressure — Baseline and follow-up examination of echocardiography is to be performed on study subjects.

SUMMARY:
This prospective study intends to explore the change of cardiac structure and function in the cohort of overweight or obesity patients, and determine the impact of clinical characteristics on cardiac remodeling and mechanics.

DETAILED DESCRIPTION:
Obesity significantly increases the risk for heart failure. Early detection of preclinical cardiac dysfunction in overweight or obesity and understanding its association with insulin resistance are of great importance.Recently, a novel technique for myocardial work (MW) assessment has been introduced to evaluate myocardial performance. To date, change of MW has been described in several cardiac conditions including dilated cardiomyopathy, significant coronary arterial diseases, and hypertrophic cardiomyopathy, which implies regional or global myocardial dysfunction. In this study, we aimed to explore the alteration of MW in overweight or obese adults and to determine whether insulin resistance or other clinical risk factors may impact myocardial mechanics before impairment of systolic function.

ELIGIBILITY:
Inclusion Criteria:

* All patients were older than 18 without any cardiac symptoms.
* The diagnosis of overweight was established when body mass index (BMI) of 25 to 30 kg/m2.
* Obese was defined as a BMI of 30 kg/m2 or higher.

Exclusion Criteria:

* diagnosis of type 2-Diabetes Mellitus according to the American Diabetes Association criteria;
* left ventricular ejection fraction<50% on echocardiography;
* arrythmia on electrocardiogram;
* severe valvular stenosis or regurgitation;
* history of coronary disease (defined as stenosis>50%) or myocardial infarction;
* stress induced wall motion abnormality on echocardiography, coronary artery stenosis >50% on coronary CT or angiography with Framingham risk score of >10;
* pacemaker or defibrillator implantation;
* the presence of bundle branch block;
* severe infection or renal dysfunction with an estimated glomerular filtration rate < 60 ml/min/1.73 m2);
* inadequate image quality on echocardiography.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: overweight or obese subjects referred to the endocrinology inpatients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
investigate the change of global myocardial work index (GWI) in overweight or obese patients | within 24 hours of the recruitment
  GWI derived from echocardiography will be assessed in overweight or obese patients and compare with lean controls
investigate the change of global constructive work (GCW) in overweight or obese patients | within 24 hours of the recruitment
  GCW will be assessed in overweight or obese patients and compare with lean controls
investigate the change of global waste work (GWW) in overweight or obese patients | within 24 hours of the recruitment
  GWW will be assessed in overweight or obese patients and compare with lean controls
investigate the change of global work efficiency (GWE) in overweight or obese patients | within 24 hours of the recruitment
  GWE will be assessed in overweight or obese patients and compare with lean controls

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China